CLINICAL TRIAL: NCT07360535
Title: Effect of Probiotic on Gut Microbiota in Young Children With Functional Constipation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Min-Tze LIONG (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Min-Tze LIONG, Prof., Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2018-027
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Functional Constipation in Children
Keywords: Bifidobacterium longum subsp. longum Dipro-X; functional constipation; infants; toddlers; probiotic
MeSH Terms: interventions — Probiotics; Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic (Experimental): Daily 6-drops of Bifidobacterium longum subsp. longum Dipro-X in non-GMO corn starch as excipient, in medium-chain triglyceride oil (1 × 10^9 CFU/day)
  Interventions: Dietary Supplement: Probiotic
- Lactulose (Active Comparator): Lactulose liquid (each 1ml contains 0.667g lactulose) 5ml/time, once a day
  Interventions: Dietary Supplement: Lactulose Oral Liquid Product
- Probiotic+Lactulose (Active Comparator): Daily 6-drops of Bifidobacterium longum subsp. longum Dipro-X in non-GMO corn starch as excipient, in medium-chain triglyceride oil (1 × 10^9 CFU/day), plus Lactulose liquid (each 1ml contains 0.667g lactulose) 5ml/time, once a day
  Interventions: Dietary Supplement: probiotic + lactulose

INTERVENTIONS:
Dietary Supplement: Probiotic — Daily 6-drops of Bifidobacterium longum subsp. longum Dipro-X in non-GMO corn starch as excipient, in medium-chain triglyceride oil (1× 10^9 CFU/day)
  Arms: Probiotic
Dietary Supplement: Lactulose Oral Liquid Product — Lactulose liquid (each 1ml contains 0.667g lactulose) 5ml/time, once a day
  Arms: Lactulose
Dietary Supplement: probiotic + lactulose — Daily 6-drops of Bifidobacterium longum subsp. longum Dipro-X in non-GMO corn starch as excipient, in medium-chain triglyceride oil (1× 10^9 CFU/day), plus Lactulose liquid (each 1ml contains 0.667g lactulose) 5ml/time, once a day
  Arms: Probiotic+Lactulose

SUMMARY:
This study was a 28-day, open-label, randomized controlled trial involving infants and toddlers diagnosed with functional constipation. Participants were randomized to receive either Bifidobacterium longum subsp. longum Dipro-X, lactulose, or a combination of both. The primary clinical outcomes assessed were bowel movement frequency, stool consistency, and defecation difficulty. To investigate potential mechanisms, stool samples were collected pre- and post-intervention for 16S rRNA gene sequencing to analyze changes in gut microbiota composition and identify specific bacterial taxa associated with clinical improvements.

DETAILED DESCRIPTION:
Functional constipation is a prevalent chronic gastrointestinal disorder with significant implications for pediatric health. Within the first year of life, many infants are affected, a figure that rises to over 10% annually. This condition not only diminishes the quality of life for infants and toddlers but also contributes to substantial healthcare costs. Early intervention is widely recognized as critical for improving treatment outcomes, underscoring the need for effective therapeutic strategies.

Growing evidence indicates that intestinal microbiota dysbiosis plays a key role in the pathogenesis of functional constipation. Studies have consistently reported reduced abundances of beneficial bacteria such as Lactobacillus and Bifidobacterium in affected individuals compared to healthy controls. These findings have spurred interest in microbiota-targeted interventions, particularly the use of Bifidobacterium, for managing constipation. Although current evidence-based guidelines do not uniformly recommend probiotics for infant constipation due to limited clinical data, their potential to restore microbial balance remains promising. Advances in genomic technologies have enabled more detailed investigations into strain-specific mechanisms, shifts in signature microorganisms, and associated symptomatic improvements, findings that may help bridge existing evidence gaps. While preclinical studies, such as those involving murine models, have shown that Bifidobacterium longum can alleviate constipation by enhancing intestinal barrier function, clinical evidence in pediatric populations remains scarce.

To address this, the present study was conducted as a randomized, open-label, three-arm controlled clinical trial. It aimed to evaluate the efficacy of Bifidobacterium longum subsp. longum Dipro-X, lactulose, and their combination in infants and toddlers with functional constipation. The study specifically assessed the intervention's effects on clinical symptoms, including defecation frequency and stool characteristics, and explored correlations between gut microbiota changes and symptom improvement. The results are intended to support the development of evidence-based, targeted microbial interventions for functional constipation in early childhood.

ELIGIBILITY:
Inclusion Criteria:

* According to the diagnostic criteria of Rome IV, the following symptoms include at least 2 and last for at least 1 month:

  1. Defecation <= 2 times per week;
  2. have a history of fecal retention;
  3. There is a history of pain or difficulty in defecation;
  4. There is a history of expelling large pieces of feces;
  5. There is a large fecal mass in the rectum. At least 1 episode of incontinence per week after self-control of bowel movements; passing large pieces of stool that may clog the toilet;
* Term infants, gestational age from 37 to 42 weeks;
* Birth weight between 2500 - 4000g;
* 0-3 years old;
* Parents voluntarily defer major changes in infant feeding practices;
* Parents are willing and able to fill in diaries and questionnaires

Exclusion Criteria:

* Chronic diseases or major medical problems;
* Gastrointestinal organic diseases;
* Growth retardation;
* The mother or child of the breastfeeding child used antibiotics within 2 weeks before randomization and during the trial;
* Infants (in formula and/or supplements) or their mothers used probiotics within 2 weeks before randomization and during the trial;
* Has participated in other clinical trials;
* Food allergies cause constipation (such as milk, eggs and other foods)

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Defecation difficulty in young children upon administration of probiotic, lactulose or their combinations as assessed via Visual Anologue Scale (VAS) | 14 days, 28 days
  Differences in defecation difficulty in young children upon administration of probiotic, lactulose or their combinations, where higher scores indicate greater defecation difficulty (worse outcome).
Bowel movement frequency in young children upon administration of probiotic, lactulose or their combinations as assessed via patients' diary | 14 days, 28 days
  Differences in bowel movement frequency in young children upon administration of probiotic, lactulose or their combinations
Bristol stool score in young children upon administration of probiotic, lactulose or their combinations as assessed via Bristol stool chart | 14 days, 28 days
  Differences in Bristol stool score in young children upon administration of probiotic, lactulose or their combinations, where lower scores indicate constipation-like outcomes and higher scores indicate diarrea-like outcomes

SECONDARY OUTCOMES:
Microbiota profiles of fecal samples in young children upon administration of probiotic, lactulose or their combinations as assessed via 16s rRNA gene sequencing | 14 days, 28 days
  Differences in microbiota profiles in fecal sample of young children upon administration probiotic, lactulose or their combinations

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, MD., Principal Investigator — Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China
Locations (2):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China
- Universiti Sains Malaysia, George Town, Malaysia

IPD SHARING:
Plan to Share IPD: No